CLINICAL TRIAL: NCT05055271
Title: Differential Diagnosis and Management of Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea: A Modified Delphi Consensus Panel Report
Brief Title: Delphi Consensus Excessive Daytime Sleepiness in OSA
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Professor Joerg Steier, Professor of Respiratory and Sleep Medicine, King's College London
Other Study IDs: 2021 EDS in OSA Delphi V1.0
Record Dates: First submitted 2021-09-07; First posted 2021-09-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; excessive daytime sleepiness; Delphi consensus
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi panel: The Delphi panel will include 10 international experts in sleep and respiratory medicine. Two panelists will serve as co-chairs and eight panelists will serve as section leads for the major topic areas throughout the process. A series of planning sessions will be conducted with the co-chairs and section leads prior to implementation of the survey.

SUMMARY:
The objective of this study is to generate expert consensus statements on the differential diagnosis, definition, and management of EDS in patients with OSA who are adequately treated with primary therapy.

DETAILED DESCRIPTION:
A study will be performed using a modified Delphi process with an international expert panel to generate recommendation statements related to the differential diagnosis and management of patients with residual EDS in OSA (and relevant sub-topics) and to determine the level of agreement for each statement from the panel as a whole. The following topics will be covered:

1. EDS: definition, evaluation/assessment, and tools
2. Definitions of residual EDS in patients with OSA treated with primary OSA therapy
3. Practical recommendations
4. Management Consensus is achieved through iterative rounds of survey and revision to the statements until a pre-determined level of agreement is met (80% agreement).

Part 1: planning and evidence review

* Series of planning sessions with co-chairs and faculty leads
* Literature is reviewed/summarized
* Initial statements will be developed based on evidence Recommendation statements on EDS in OSA will be formulated and rated according to level of agreement on a 5-point Likert scale.

Part 2: Survey to achieve consensus

* Survey, based on the initial statements developed by faculty leads, will be developed to allow for vetting by full faculty group
* At least 3 rounds of review (2 remote and 1 live [virtual]) will be held to achieve consensus on each topic of interest and finalize consensus statements

ELIGIBILITY:
Inclusion Criteria:

* Members of the panel include experts in sleep and respiratory medicine in North American and Europe.

Exclusion Criteria:

* Panelists who were not able to commit to all rounds of the modified Delphi process will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experts in sleep and respiratory medicine from North America and Europe
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Consensus | 6 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating a given statement A+ or A.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, PhD, Study Chair — King's College London (KCL), UK; Atul Malhotra, MD, Study Chair — University of California San Diego (UCSD), USA
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Background] Rosenberg R, Schweitzer PK, Steier J, Pepin JL. Residual excessive daytime sleepiness in patients treated for obstructive sleep apnea: guidance for assessment, diagnosis, and management. Postgrad Med. 2021 Sep;133(7):772-783. doi: 10.1080/00325481.2021.1948305. Epub 2021 Jul 22. PMID 34292843